CLINICAL TRIAL: NCT06492356
Title: Impact of Tripolar Radiofrequency on Acne Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alshymaa Ahmed Kamel Ahmed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alshymaa M.sc
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic; Scar; Radiofrequency
MeSH Terms: conditions — Hypertrophy; Cicatrix

STUDY DESIGN:
Intervention Model Description: single-blinded randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Consists of 20 patients with acne scars and will receive medical treatment by a dermatologist and tripolar radiofrequency (RF) therapy once a week for 12 weeks, each session for 15 minutes.
  Interventions: Device: Tripolar radiofrequency therapy; Drug: medical treatment
- Group B (Active Comparator): consists of 20 patients with acne scars and will receive medical treatment by a dermatologist
  Interventions: Drug: medical treatment

INTERVENTIONS:
Device: Tripolar radiofrequency therapy — Twenty patients underwent weekly TriPollar RF treatment, using a new RF technology with three or more electrodes. Glycerin was applied to the treatment area before and after each session, with the procedure lasting 15 minutes. The technology uses a sequence of electrical modulation to prevent overheating and requires no active cooling of the electrodes or skin.
  Arms: Group A
Drug: medical treatment — Twenty patients will receive medical treatment by dermatologist.

SUMMARY:
The aim of this study is to investigate the therapeutic efficacy of tripolar radiofrequency on acne scar

DETAILED DESCRIPTION:
Acne scarring is a very troublesome complication associated with acne and is reported in as high as 95% of the patients, sometimes even with proper and prompt treatment. The visible depressed scars have been known to have a negative impact on patient's psychological well-being and quality of life. Post acne scarring can pose as a risk factor for depression, anxiety, and even suicide (Villani, 2020).

There are a multitude of treatment options that are traditionally used for the treatment of acne scars including many ablative and non-ablative methods (Dogra, 2014).

Furth more, the need of this study is developed from the lack in quantitative knowledge and information in the published studies which investigate the effect of tripollar RF This study will be designed to provide guidelines about the effect tripollar Radiofrequency on acne scars.

ELIGIBILITY:
Inclusion Criteria:

* Forty patients having acne scar, from both genders their ages will be ranged from 20 to 40 years old
* Both genders will participate in this study as the following distribution 17 male and 23 female.
* They diagnosed as acne scar by their physicians and referred for physical therapy management.
* Medically and psychologically stable patients.
* All patients will approve and sign a consent form before starting the program which will include the purpose, natures and potential risks of the study which will be explained to all patients

Exclusion Criteria:

* Patients who suffer from hypertrophic and/or keloidal scars and a skin condition in the area of acne scars that would interfere with study procedures (e.g., plaque psoriasis, tattoo, birthmark, facial hair).
* Patients with medical red flags as severe psychiatric disorder or cognitive deficits.
* Medically unstable and uncooperative patients.
* Untreated and active/ongoing acne vulgaris.
* Immunocompromised status.
* History of skin cancer.
* Recurrent herpes viral infection.
* Pregnancy or breastfeeding status.
* Females take contraceptive pills
* Hormonal disturbance

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Assessing the change in severity of acne scars | at base line and following 12 weeks
  SCARS is a 5-item instrument designed to rate the severity of acne scars in a mirror. It uses visual analog scales to differentiate between active and scars. The tool is self-completion and can be completed quickly. Patients are photographed at the beginning and after 12 treatment sessions. SCARS scores range from 0 to 4, with higher scores indicating greater severity. It captures demographic information and clinical characteristics of acne and scarring.

SECONDARY OUTCOMES:
Assessing the quantitative measurement of the acne scars | at base line and following 12 weeks
  Dey et al. developed an automatic approach to quantify acne scars using color images, achieving a sensitivity of 90.36 and specificity of 93.82. However, this method does not allow for volumetric assessment of the scar. Another technique, proposed by Petukhova et al., uses three-dimensional photographic images to construct a topographic map, which is then objectively calculated for each scar. This method does not assess color changes like dyspigmentation, which is essential for tracking scars over time. Further testing is needed to improve this method.

CONTACTS AND LOCATIONS:
Locations (1):
- Malawy Specialized Hospital, Minya, Egypt